CLINICAL TRIAL: NCT06010576
Title: Endoscopic Ultrasound-guided Rendezvous Technique Versus Early Precut Papillotomy for Difficult Bile Duct Cannulation During Endoscopic Retrograde Cholangiopancreatography: a Multicenter Randomized Controlled Trial
Brief Title: Endoscopic Ultrasound-guided Rendezvous Versus Precut Papillotomy
Acronym: ERVPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tokyo University (Other); Gifu University Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Assitant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.720-T
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Bile Duct Diseases
Keywords: ERCP, EUS
MeSH Terms: conditions — Bile Duct Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided rendezvous group (EUS RV group) (Active Comparator): In the EUS RV group, a linear array echoendoscope would be used to evaluate the common bile duct and left intrahepatic duct in order to identify the optimal route for biliary access by fine needle. Using a 19 gauge EUS needle, the dilated biliary tree will be accessed by either a transduodenal puncture to the common bile duct or a transgastric puncture to the left intrahepatic duct under direct EUS guidance. The optimal access route will be based on patient's anatomy after EUS assessment and left to the discretion of the investigator. Next, a guidewire would be advanced through the needle into the bile duct and out of the papillary orifice. The echoendoscope would then be exchanged to a duodenoscope for ERCP. The EUS rendezvous ERCP procedure will be completed by retrieving the rendezvous guidewire into the duodenoscope or by cannulation alongside the rendezvous guidewire to obtain biliary access.
  Interventions: Procedure: EUS-guided rendezvous
- Early precut papillotomy group (EPP group) (Active Comparator): In the EPP group, the precut papillotomy would be performed with 1 of the following acceptable techniques per the usual practice of the study investigator and institution: 1) conventional precut papillotomy by needle knife, 2) precut fistulotomy by needle knife, or 3) transpancreatic precut papillotomy by papillotome
  Interventions: Procedure: Early precut papillotomy group

INTERVENTIONS:
Procedure: EUS-guided rendezvous — A linear array echoendoscope would be used to evaluate the common bile duct and left intrahepatic duct in order to identify the optimal route for biliary access by fine needle. Using a 19 gauge EUS needle, the dilated biliary tree will be accessed by either a transduodenal puncture to the common bile duct or a transgastric puncture to the left intrahepatic duct under direct EUS guidance. The optimal access route will be based on patient's anatomy after EUS assessment and left to the discretion of the investigator. Next, a guidewire would be advanced through the needle into the bile duct and out of the papillary orifice. The echoendoscope would then be exchanged to a duodenoscope for ERCP. The EUS rendezvous ERCP procedure will be completed by retrieving the rendezvous guidewire into the duodenoscope or by cannulation alongside the rendezvous guidewire to obtain biliary access.
  Arms: EUS-guided rendezvous group (EUS RV group)
Procedure: Early precut papillotomy group — The precut papillotomy would be performed with 1 of the following acceptable techniques per the usual practice of the study investigator and institution: 1) conventional precut papillotomy by needle knife, 2) precut fistulotomy by needle knife, or 3) transpancreatic precut papillotomy by papillotome
  Arms: Early precut papillotomy group (EPP group)

SUMMARY:
Selective bile duct cannulation is the most important step in endoscopic retrograde cholangiopancreatography (ERCP) for treatment of benign and malignant pancreatobiliary diseases, but it may fail in up to 15% of cases. Precut papillotomy is an advanced ERCP cannulation technique recommended by guidelines for rescue of difficult biliary access, but it is not without limitations. Endoscopic ultrasound (EUS)-guided biliary drainage is a novel interventional EUS technique that has been increasingly performed after failed biliary access by advanced ERCP cannulation techniques.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is the preferred therapeutic modality over surgery or interventional radiology procedures in many common benign or malignant pancreatobiliary diseases in modern clinical practice, but selective bile duct cannulation may fail in up to 15% of cases.

The implication of failed endoscopic biliary access can be substantial for the following reasons: higher risk of post-ERCP pancreatitis (PEP), need for rescue procedures such as external biliary drainage by interventional radiology, risks of external biliary drainage catheter-related complications including catheter blockage.

Advanced ERCP cannulation techniques such as pancreatic guidewire-assisted biliary cannulation with or without pancreatic stenting, and precut papillotomy are recommended by guidelines in patients with difficult bile duct cannulation, but they are not without limitations. If pancreatic duct cannulation is not feasible or pancreatic guidewire-assisted biliary cannulation fails, precut papillotomy using 1 of the 3 accepted precut techniques: 1) conventional precut papillotomy by needle knife, 2) precut fistulotomy by needle knife, or 3) transpancreatic precut papillotomy by papillotome, can be performed depending on institutional expertise. Despite a higher biliary cannulation success by precut papillotomy when compared to pancreatic guidewire-assisted biliary cannulation, a higher risk of PEP has also been traditionally associated with precut papillotomy when it is performed after prolonged cannulation attempts. On the other hand, there has been growing evidence to suggest the increased risk of PEP may be related to the persistent cannulation attempts before precut rather than the precut papillotomy itself. In a recent meta-analysis of 5 randomized controlled trials comparing "early precut papillotomy" to persistent standard cannulation techniques in ERCP by attending endoscopists and advanced endoscopy trainees, the incidence of PEP was not significantly different between the "early precut papillotomy" and the persistent standard cannulation groups.

EUS-guided rendezvous technique (EUS RV) is a novel advanced interventional EUS technique that has been increasingly performed in tertiary centers for patients with failed biliary access by advanced ERCP cannulation techniques. Several variations of EUS-guided biliary drainage procedures have been described including transpapillary drainage procedures (EUS RV for biliary access, EUS-guided antegrade stenting) and transmural drainage procedures (EUS-guided choledochoduodenostomy, EUS-guided hepaticogastrostomy). EUS RV can be applied in both benign and malignant biliary conditions as a salvage technique for difficult biliary access when the major papilla is accessible. EUS RV involves the following key steps: access of the dilated bile duct by a EUS needle under EUS guidance, performance of cholangiogram, advancement of the rendezvous guidewire into the bile duct and out of the major papilla into duodenum, and exchange of echoendoscope back to a duodenoscope to complete the procedure by retrieving the rendezvous guidewire into the duodenoscope or by cannulation alongside the rendezvous guidewire. Because EUS RV achieves biliary access by targeting the dilated bile duct with antegrade passage of guidewire from bile duct through the papillary orifice, theoretically this would carry a lower risk of procedure-related PEP when compared to early precut papillotomy.

In a recently published consensus guidelines on the optimal management in interventional EUS procedures proposed by experts from our endoscopy research group and other member institutions of the Asian EUS Group, EUS-guided biliary drainage is recommended as the procedure of choice for biliary drainage in patients with failed ERCP when expertise is available based on high level evidence. The technical success of EUS RV has increased over time to 73% to 100% in studies published after 2012.

Studies directly comparing EUS RV and precut papillotomy in patients with difficult biliary access remain scarce. In a single center retrospective study published in 2012 comparing the clinical outcomes of 58 EUS RV procedures and 144 precut papillotomy procedures in patients with failed bile duct cannulation in ERCP, Dhir V et al reported a significantly higher first session technical success of biliary access (98% vs 90%, p = 0.038) and a lower adverse event rate (3.4% vs 6.9%, p = 0.27) in the EUS RV group. In a multicenter retrospective study published in 2017 by Lee A et al comparing the clinical outcomes of 50 EUS RV + 11 EUS-guided transmural drainage procedures and 142 precut papillotomy procedures in patients with failed bile duct cannulation in ERCP, a higher technical success of biliary access (94% vs 75%) was also demonstrated in the EUS RV group.

Despite the promising results of EUS RV in patients with failed biliary cannulation by advanced ERCP techniques, there has been no dedicated randomized controlled trial directly comparing EUS RV and early precut papillotomy in patients with difficult bile duct cannulation. We aim to conduct a multicenter randomized controlled trial comparing the clinical efficacy of these 2 advanced endoscopic biliary access techniques in patients with difficult bile duct cannulation in ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older undergoing ERCP with indication for bile duct cannulation
* Native major papilla
* Difficult bile duct cannulation, defined by the presence of 1 of the following: 1) unsuccessful bile duct cannulation within 10 cannulation attempts, 2) unsuccessful bile duct cannulation within 10 minutes spent in cannulation, or 3) 2 unintended pancreatic duct cannulation or opacification with contrast
* Written informed consent available

Exclusion Criteria:

* Unable to provide written informed consent
* Contraindications for endoscopy due to comorbidities
* Prior biliary sphincterotomy
* Surgically altered upper gastrointestinal anatomy or duodenal obstruction precluding a standard ERCP
* Uncorrectable coagulopathy (INR > 1.5) and thrombocytopenia (platelet < 50,000) by blood product transfusion
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The first session technical success for biliary access by EUS-guided rendezvous technique and early precut papillotomy in patients with difficult biliary access during ERCP | Intra-procedure, during ERCP
  Technical success by EUS RV is defined as successful EUS-guided needle access of bile duct confirmed by bile aspiration and cholangiogram, advancement of guidewire into bile duct and out of papilla, and obtaining deep biliary cannulation by retrieving the rendezvous guidewire into duodenoscope or by cannulation alongside the rendezvous guidewire. Technical success by Early Precut Papillotomy is defined as successful bile duct access by 1 of the 3 acceptable precut techniques in achieving deep biliary cannulation, confirmed by bile aspiration and cholangiogram.

SECONDARY OUTCOMES:
Procedure-related serious adverse events in the EUS-guided rendezvous group and the early precut papillotomy group within 30 days of ERCP | From day of procedure to Day 30 after procedure
  Procedure-related serious adverse events include perforation, bleeding, biliary sepsis, pancreatitis, bile leak, or procedure-related mortality
Procedure time to achieve biliary access by the assigned study biliary access technique | Intra-procedure, during ERCP
  EUS RV group: time from EUS-guided needle access of bile duct to successful biliary cannulation by ERCP. Early Precut Papillotomy group: time from precut initiation to successful biliary cannulation.
Need for rescue biliary drainage procedures in patients with failed biliary access by the assigned study technique, including crossover to the other study biliary access technique, need for PTBD by interventional radiology | Intra-procedure (during ERCP) and 3 days post procedure
  Intra-procedure: crossover to the other study biliary access technique. Within 3 days of procedure: need for percutaneous transhepatic biliary drainage by interventional radiology

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tang, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No